CLINICAL TRIAL: NCT07049809
Title: Targeting Sarcopenia and Frailty: Multicomponent Exercise With Focal Muscle Vibration to Reduce Sarcopenia, Frailty Levels, and Cognitive Impairment in Institutionalized Older Adults
Brief Title: Targeting Sarcopenia and Frailty: Multicomponent Exercise With Focal Muscle Vibration
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitat Internacional de Catalunya (Other)
Responsible Party: Principal Investigator, Sergi Rodriguez Rodriguez, Physiotherapist. Professor at the department of Medicine., Universitat Internacional de Catalunya
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 01-24-175-116
Record Dates: First submitted 2025-06-25; First posted 2025-07-03 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-07

CONDITIONS: Sarcopenia; Frailty at Older Adults; Cognitive Impairment; Adherence
Keywords: sarcopenia; frailty; older adults; cognition; focal vibration; multicomponent exercise
MeSH Terms: conditions — Sarcopenia; Cognitive Dysfunction; Frailty

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Combination Intervention group (Experimental): 2-month intervention. 3 days/week. 30 minutes/day. Will receive a multicomponent program based on aerobic training, resistance training and balance training, combined with focal muscle vibration. Of the 3 days of weekly intervention, 1 day will be aerobic exercise combined with focal muscle vibration, 1 day resistance exercise with focal muscle vibration and 1 day of balance exercise with focal muscle vibration.
  The combined program will be individualized based in the intrinsic capabilities of each individual.
  Interventions: Combination Product: Focal Muscle Vibration; Other: Multicomponent Exercise
- Multicomponent Exercise Group (Active Comparator): 3-month intervention. 3 days/week. 30 minutes/day. Will receive a multicomponent program based on aerobic training, resistance training and balance training.
  The combined program will be individualized based in the intrinsic capabilities of each individual.
  Interventions: Other: Multicomponent Exercise

INTERVENTIONS:
Combination Product: Focal Muscle Vibration — The focal vibration machine will be used. The device has 6 muted transducers that generate power between 30-300 Hz, but for this study we will use between 100-150 Hz for 30 minutes.
  The application of the 6 transducers or heads is at the level of the lower extremities, since those muscle groups present the most clinical correlation with functional parameters such as gait and balance. 3 transducers will be placed on one leg (vastus medialis, vastus lateralis and rector anterior) and the other 3 transducers on the other leg, on the same muscles. To speed up the intervention program and cover more participants, 4 focal vibration machines will be used. Each participant wil use 1 machine and 6 transducers, so during the 30 minutes that the intervention lasted, the groups will be of 4 participants with t
  Arms: Combination Intervention group
Other: Multicomponent Exercise — The program consists of a multi-component approach, integrating aerobics, resistance, and balance training. The weekly schedule include three intervention days: one day focused on aerobic exercise, one day dedicated to resistance training and one day centered on balance training. The combined program is individualized based on the intrinsic capabilities of each individual.

SUMMARY:
This study aimed to evaluate the efficacy of multicomponent exercises (aerobic exercises, strength exercises, and balance exercises), individualized with the application of a focal muscle vibration machine at the lower extremities, on parameters of sarcopenia (a muscle disease) in health-related physical fitness, physical performance, frailty levels, and cognitive function, falls, and hospitalizations in older adults.

Focal muscle vibration is a type of therapeutic technique used with the application of six capsules placed on the lower extremities, three on each bed, each of which generates a tolerable vibration depending on the stimulation of the muscles. It is neither painful nor counterproductive to the muscles in the lower extremities.

Multicomponent exercises refer to the application of exercises through three different modalities: aerobic exercises, strength exercises, and balance exercises. We alternate these three types of exercises to achieve millions of health benefits. The multi-component program will be individualized based on each individual's abilities to avoid risks and achieve maximum benefits.

DETAILED DESCRIPTION:
This study presents the hypothesis that it will allow researchers to significantly improve health parameters in very fragile people, which may have positive impacts at both the individual and community levels. The incorporation of focal vibration as part of a multicomponent approach to exercise is innovative and opens new lines of research in the field of rehabilitation and developmental health. Currently, I understand that there is a growing need to address the healthy development and fragility of the large adult population, given the increasing proportion in today's society and the reptes associated with the loss of functional abilities, which studies can allow other scientists to see the benefits of the program in different areas. health parameters after 3 months of intervention.

The participation in the study will include:

* Authorizing the investigators to access your medical history. This will allow the investigators to collect information about the clinical data of the participants.
* Authorizing the investigators to share coded clinical information with other research teams. Theparticipant authorize access to information related to hospitalizations and drugs consumed.
* Allow the collection of data both at the beginning and after the intervention after 3 months by the external research team. Different data will be collected in a single day both at the beginning and at the end of the intervention, with an approximate duration of 35/40 minutes per person. The data that will be collected will give the researchers information about functional status, muscle strength and power and cognitive level. In addition. the levels of sarcopenia in dominant leg will be evaluated with ultrasound. The ultrasound assessment is a painless test through which an attempt will be made to see the amount of muscle and fat present at the level of the dominant lower extremity. In addition, at the beginning and end of the intervention a blood test will be performed by CST personnel. This analysis will be used to evaluate different blood markers of the participants and see how they respond to the different intervention programs.
* Randomization to one of the 2 study groups: a focal vibration group with multicomponent exercise, an exercise only group.

Prior to the start of the intervention program, and after this 3-month period, a series of functional tests, tests, muscle ultrasound and a blood analysis will be performed. These tests are tests that are normally used in clinics or hospitals as functional or force assessments in the geriatric population. Once the initial evaluation and data analysis has been carried out, a group will subsequently be randomly assigned to one of the 3 groups that is proposed by the study. If still assigned to group 1) combined exercise with focal vibration, repeat for 3 months, 3 days per week and 30 minutes per day, multicomponent exercises (strength, aerobic exercise and balance) combined with focal muscular vibration. In case it continued to be assigned to group 2) multicomponent exercise, repeat for 3 months, 3 days per week and 30 minutes a day, multicomponent exercises (strength, aerobic exercise and balance).

ELIGIBILITY:
Inclusion Criteria:

* people over 75 years of age,
* score ≥18 on the Mini-Mental State Exam (MMSE)
* score on the Clinical Frailty Scale between 1-6
* be institutionalized
* ability to sit unassisted on a chair or in a wheelchair

Exclusion Criteria:

* progressive degenerative diseases
* uncontrolled symptomatic cardiovascular or respiratory disease
* current cancer under treatment
* severe audiovisual impairment

Min Age: 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-07-02 (Estimated); Primary Completion 2025-09 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Short Physical Performance Battery | From enrollment to the end of treatment at 12 weeks
  Short Physical Performance Battery (SPPB) is a standardized test that evaluates Balance, Gait speed and Lower limb strength (via chair stands). Has a total puntuaction of 12 points: 0-3: Severe physical limitation, 4-6: Moderate limitation, 7-9: Mild limitation, 10-12: Good physical function. The SPPB (Short Physical Performance Battery) is closely related to sarcopenia because it assesses physical function, which is one of the key diagnostic criteria for sarcopenia.

SECONDARY OUTCOMES:
Demographic and anthropometric assessments | from enrollment to 12 weeks after treatment
  Age, height, and weight will be provided by the residence physiotherapist with the data they previously had with the clinical histories. BMI will be calculated using the formula BMI = kg/m2. We will use the WHO recommendations for adult population to obtain the categories of "individuals with obesity and without obesity": a) BMI < 30: without obesity and b) BMI ≥ 30: with obesity. The length of time each participant has been institutionalized in the residence will also be taken into account.
Handgrip | from enrollment to 12 weeks after intervention
  Handgrip strength will be assessed with the Jamar hand dynamometer (Sammons Preston, Inc., Bolingbrook, IL, USA) in kilograms. Participants will be seated with their elbows flexed at 90° and performing a maximal handgrip strength for three seconds three times with each hand. The mean of the three attempts on each arm will be used in the analysis. This procedure has been shown to have excellent reliability (ICC = 0.85-0.98). Cutoffs are a low handgrip strength of less than 27 kg for men and less than 16 kg for women.
SARC-F | from enrollment to 12 weeks after intervention.
  SARC-F is a simple, fast screening questionnaire used to identify people at risk of sarcopenia. The SARC-F scale includes 5 components: strength, walking assistance, getting up from a chair, climbing stairs, and falls. Scores range from 0 to 10, with 0 to 2 points for each component. A SARC-F score ≥ 4 suggests a high risk of sarcopenia and signals the need for further assessment (e.g., grip strength, SPPB, muscle mass)
Clinical Frailty Scale | from enrollment to 12 weeks after intervention
  The Clinical frailty scale (CFS) evaluates specific domains including comorbidity, function, and cognition to generate a frailty score ranging from 1 (very fit) to 9 (terminally ill). Frailty will be assessed using this scale at the beginning before the intervention and after 6 months, at the end of the program. CFS degrees 1-4 denote non-frailty (declining degrees of robustness), whereas degrees ≥5 indicate frailty
Muscle ultrasound | from enrollment to 12 weeks after intervention.
  Muscle thickness and cross-sectional area of the rectus femoris, quadriceps and vastus lateralis will be assessed before the intervention and after 3 months . VScan pocket-sized ultrasound with dual probe (GE Healthcare, United States) will be used. The linear probe provides a 2.9 cm aperture and works across a frequency range of 3.4 to 8.0 MHz. For rectus femoris imaging, the depth of imaging will be adjusted until the femur is visualized, and the rectus femoris could be seen superior to vastus intermedius. The probe will be placed perpendicular to the long axis of the femoral shaft. For vastus lateralis visualization, the probe will be placed parallel to the long axis of the femoral shaft, and the depth of imaging will be adjusted until the deep aponeurosis of the vastus lateralis, and the vastus intermedius inferior to it, could be visualized. A large amount of water-based gel will be used, and minimal pressure will be placed on the probe to prevent compression of muscle.
Mini Mental State Exam | from enrollment to 12 weeks after intervention.
  The MMSE evaluates several cognitive domains, including orientation, registration, attention and calculation, short-term memory (recall), language, and visuospatial abilities. During the assessment, individuals are asked to perform tasks such as identifying the current date and location, repeating and later recalling a set of words, performing basic arithmetic (e.g., serial sevens), naming objects, following written and verbal commands, writing a sentence, and copying a geometric figure.
  The total MMSE score ranges from 0 to 30 points. Higher scores indicate better cognitive function.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Cordes T, Bischoff LL, Schoene D, Schott N, Voelcker-Rehage C, Meixner C, Appelles LM, Bebenek M, Berwinkel A, Hildebrand C, Jollenbeck T, Johnen B, Kemmler W, Klotzbier T, Korbus H, Rudisch J, Vogt L, Weigelt M, Wittelsberger R, Zwingmann K, Wollesen B. A multicomponent exercise intervention to improve physical functioning, cognition and psychosocial well-being in elderly nursing home residents: a study protocol of a randomized controlled trial in the PROCARE (prevention and occupational health in long-term care) project. BMC Geriatr. 2019 Dec 23;19(1):369. doi: 10.1186/s12877-019-1386-6. PMID 31870314
- [Background] Cruz-Jentoft AJ, Bahat G, Bauer J, Boirie Y, Bruyere O, Cederholm T, Cooper C, Landi F, Rolland Y, Sayer AA, Schneider SM, Sieber CC, Topinkova E, Vandewoude M, Visser M, Zamboni M; Writing Group for the European Working Group on Sarcopenia in Older People 2 (EWGSOP2), and the Extended Group for EWGSOP2. Sarcopenia: revised European consensus on definition and diagnosis. Age Ageing. 2019 Jan 1;48(1):16-31. doi: 10.1093/ageing/afy169. PMID 30312372